CLINICAL TRIAL: NCT06789666
Title: Feasibility of a Digital Art Therapy Application Designed to Improve Quality of Life in Young Cancer Survivors
Brief Title: Digital Art Therapy for Young Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Ian's Friends Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC2339
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Pediatric Cancer; Pediatric Malignancies; Pediatric Sarcoma of Soft Tissue; Adolescent and Young Adult With Brain Cancer
Keywords: therapy; art; mental health quality of life; patient-reported outcome; ARTCan application; digital art therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital Art Therapy (Experimental): All participants will receive art therapy via the ARTCan App for 6 weeks, and will also be prompted to complete mental health quality of life surveys at baseline and each week, which will be available for the therapist to review.
  Interventions: Behavioral: ARTCan App

INTERVENTIONS:
Behavioral: ARTCan App — The ARTCan App is an art therapy technology application program. The application can be accessed via the web (via computer, phone, or on a device such as an iPad). With the use of the application, participants complete weekly sessions that culminate in an "art" piece. Note that participants are not required to have expertise in drawing; developing art skills or assessing the quality of art pieces is not the focus of the ARTCan program.
  Subjects will upload a photo of the art they created to this application to show proof of completion of art therapy. They will also answer questions specific to the art therapy theme for the week.

SUMMARY:
This is a single-site, single-arm, interventional study assessing the feasibility of the ARTCan Therapy Application (App) and whether it is an acceptable means of administering art therapy to young adult cancer survivors. The ARTCan Therapy App guides participants through a 6-week digital art therapy program. Subjects will participate in weekly art therapy prompts guided by the app and will complete weekly mental health quality of life (MHQoL) surveys during the intervention. In addition, baseline and end-of-intervention patient-reported outcome measures (PROMIS-DSF8a) and an acceptability survey will be administered. The hypothesis is that digital art therapy is feasible for young adult cancer survivors with self-reported mood issues and is an acceptable means of administering art therapy in the patient population.

DETAILED DESCRIPTION:
The ARTCan application has been designed to define therapy strategies for the care of patients; it emerges from a unique collaboration in the disciplines of design, art, art therapy, and medicine from the College of Design, Architecture, Art, and Planning (DAAP) at the University of Cincinnati (UC) and the School of Medicine, the University of North Carolina, Chapel Hill. The relevance of the application design was to enable the trans-disciplinary team to experiment with proof of the following concepts: 1) technology-based tools and feasibility studies for new lines of research in treatment; 2) research that embraces intellectual diversity by merging the creative disciplines; and 3) addressing issues of health and well-being of patients. This study is testing whether the digital art therapy application "Art Therapy Can Do" (ARTCan) is a feasible means of administering art therapy to young cancer survivors. The study is funded by the Ian's Friends Foundation and the Weatherspoon Foundation.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study a subject must meet all of the eligibility criteria outlined below.

* Written informed assent and parental consent obtained to participate in the study and HIPAA authorization for release of personal health information.
* Subject is willing and able to comply with study procedures based on the judgment of the investigator.
* Age 18-25 years at the time of consent.
* Childhood cancer survivor, defined as having cancer between birth 17 years of age and who has completed cancer treatment.
* Reliable internet connection and access to a computer, smartphone, or iPad to support application and virtual study visits.
* Answers "yes" to the question "Do you experience mood issues (yes or no)?".

Exclusion Criteria:

* All subjects meeting any of the exclusion criteria at baseline will be excluded from study participation.
* Patients who lack interest in art. Screening question: Are you open to making art on a scale from 1-5 (1 being not at all, and 5 being very much; must score 3 or higher).
* Subjects who lack basic technology skills (Screening question: On a scale of 1-5 (1 being uncomfortable, and 5 being very comfortable), how would you rate your comfort using websites. Must score 3 or higher).
* Subjects unable to provide consent.
* Other conditions or factors which in the opinion of the Pl would not make the patient a good candidate for the study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of art therapy | Up to 6 weeks
  The feasibility of art therapy will be determined by the proportion of participants who complete art therapy. The proportion of participants who complete 4 of the 6 art therapy modules will be determined. A completion rate of 10 out of 15 participants will be deemed feasible.

SECONDARY OUTCOMES:
Acceptability of art therapy | at 6 week
  Acceptability of art therapy will be measured as the proportion of participants responded to the survey questionnaire administered at the end of the intervention. The survey questionnaire will be taken via a web-based application as post- Intervention Assessment. Question: 1) Please provide your impression of the ARTCan App: A) I like the App B) I don't like the.

CONTACTS AND LOCATIONS:
Overall Officials: Soma Sengupta, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials